CLINICAL TRIAL: NCT02047383
Title: Repercussion of Hospital Stay in Patients With Respiratory Infection
Brief Title: Hospital Stay and Respiratory Infection
Status: Completed | Type: Observational
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Marie Carmen Valenza, assistant professor, Universidad de Granada
Other Study IDs: DF0047UG
Record Dates: First submitted 2014-01-22; First posted 2014-01-28 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Respiratory Infection
Keywords: respiratory infection; physical variables
MeSH Terms: conditions — Respiratory Tract Infections | interventions — Cold Temperature

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- respiratory infection: Hospitalized patients with a respiratory infection
  Interventions: Other: Respiratory infection

INTERVENTIONS:
Other: Respiratory infection — An assessment of the patients included in the study will be conducted
  Other Names: Descriptive

SUMMARY:
The acute respiratory infection is the fourth most common cause of hospital stay between elderly people. The purpose of this study is to evaluate the repercussion of hospital stay in hospitalized patients with a respiratory infection.

DETAILED DESCRIPTION:
Acute respiratory infection is a serious infection that prevents normal breathing function. It refers to any of a number of infectious diseases involving the respiratory tract. Health conditions that increase the risk of a respiratory infection include: another lung condition, a heart condition, a kidney or liver condition and a lowered immune system. The hospital stay of this patients is approximately 7-10 days and it is important to study the effects of this stay in the physical and psycho-emotional characteristics of patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of respiratory infection
* Age: more than 50 year.
* Signed written consent.

Exclusion Criteria:

* Heart disease and concomitant neurological condition.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients with an acute respiratory infection
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2014-01; Primary Completion 2014-05 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Strength in upper and lower limbs | Participants will be followed for the duration of hospital stay, an expected average of 8 days
  The quadriceps and the hand-grip strength is assessed using a dynamometer with a standard protocol allowing three attempts on each side. During each measurement, patients were sitting with their shoulder adducted and elbow flexed to 90°. The maximum value achieved was used in the analyses. This is important in order to quantify the increase of strength Kg/cm2 The test 2-minute step in place is also going to be used for this purpose, counting the times the patients go up the right knees in two minutes.

SECONDARY OUTCOMES:
Quality of life | Participants will be followed for the duration of hospital stay, an expected average of 8 days
  The quality of life associated with health is going to be measure with t the EuroQol-5 questionnaire.
Lung function | Participants will be followed for the duration of hospital stay, an expected average of 8 days
  Lung function is going to be evaluated using a spirometer.
Activity monitoring | Participants will be followed for the duration of hospital stay, an expected average of 8 days
  The accelerometer Armband is going to be used for activity monitoring. It measures the intensity of the activity during 12 hours.
Quality of sleep | Participants will be followed for the duration of hospital stay, an expected average of 8 days
  Changes in quality of sleep. For this purpose, the participants are going to complete the Pittsburgh Quality of Sleep Index. This is a self-rating questionnaire with seven subscores that result in a global score between 0 and 21.
Mood | Participants will be followed for the duration of hospital stay, an expected average of 8 days
  Mood in these patients will be measured by the Hospital Anxiety and Depression Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Carmen Valenza, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- Faculty of health Sciences. University of Granada, Granada, Spain, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Martin-Salvador A, Torres-Sanchez I, Saez-Roca G, Lopez-Torres I, Rodriguez-Alzueta E, Valenza MC. Age group analysis of psychological, physical and functional deterioration in patients hospitalized for pneumonia. Arch Bronconeumol. 2015 Oct;51(10):496-501. doi: 10.1016/j.arbres.2014.11.009. Epub 2015 Jan 17. English, Spanish. PMID 25605525